CLINICAL TRIAL: NCT01576939
Title: A Feasibility Study of IMRT (Intensity Modulated Radiotherapy) Modulation to Account for Scattered Radiation From Dental Fillings in Head and Neck Cancer Patients
Brief Title: Feasibility of IMRT Modulation to Account for Scattered Radiation From Dental Fillings in Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Quynh-Thu Le, Professor of Radiation Oncology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-21777; SU-08102011-8266 (Other: Stanford University); ENT0032 (Other: OnCore)
Record Dates: First submitted 2011-09-23; First posted 2012-04-13 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMRT Modulation (Experimental): All patients will undergo a computed tomography (CT) simulation study +/- a positron emission tomography (PET) scan using ≤ 3mm slices for radiation treatment planning. A standard, "non-filling" optimized IMRT (Intensity Modulated Radiation Therapy) plan will be generated and patients will be treated with megavoltage radiation over a course of > 6 weeks with a planned tumor dose of > 60 Gy. A medical doctor will perform weekly mucositis evaluation and grading for the measured site once a week during radiation therapy
  Modulation of an IMRT plan to reduce the dose to less than 35 Gy delivered to adjacent normal mucosa surrounding the dental filling without compromising normal tissue or tumor doses.
  Interventions: Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Radiation: Intensity Modulated Radiation Therapy — We are using thermoluminescent dosimeter (TLD) to measure the mucosal dose adjacent to the dental fillings in a standard, "non-filling" optimized IMRT (intensity modulated radiotherapy treatment) plan that is normally delivered in the clinic. If the measured mucosal dose exceeds 35 Gy, we will generate a "filling" optimized IMRT plan to reduce it to < 35 Gy. The new plan will be deemed acceptable and implemented only if it does not (1) compromise the tumor coverage, (2) increase the dose to either the remaining oral cavity or the spared parotid gland(s).
  Other Names: IMRT

SUMMARY:
The main objective of this study is to determine the feasibility of optimizing the IMRT treatment plan based on dosimeter measurements of mucosal radiation dose adjacent to the dental fillings to reduce such dose to < 35 Gy without compromising tumor coverage and/or increasing the dose to the remaining oral cavity or nearby parotid glands.

DETAILED DESCRIPTION:
Using radiation dosimeter, we will perform measurement of the doses received by the mucosa adjacent to the dental fillings in patients receiving IMRT for head and neck cancer. If the mucosa dose is estimated to be greater than 35 Gy for the entire radiation course, we will generate and implement a "filling" optimized IMRT plan, provided that this new plan does not compromise tumor coverage or increase dose to the rest of the oral mucosa or parotid glands. Dosimeter will be used to measure the mucosal dose delivered by this new IMRT plan. Patient's mucositis grade, narcotic use and self-reported mouth and throat soreness scores will be recorded and correlated to mucosal dose. We hypothesize that modulation of an IMRT plan to reduce the dose delivered to adjacent normal mucosa surrounding the dental filling can decrease the severity and duration of radiation-related oral mucositis. Here we propose to use thermoluminescent dosimeter (TLD) to measure the mucosal dose adjacent to the dental fillings in a standard, "non-filling" optimized IMRT plan that is normally delivered in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HNC undergoing radiation therapy +/- chemotherapy at Stanford University
* At least 18 years old
* Metallic filling present
* Planned radiation dose to the tumor > 60 Gy at 1.8 to 2.2 Gy/fx
* Able to understand and sign a written informed consent document.

Exclusion Criteria:

* Pregnant
* Nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2014-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Thu Le, MD, Principal Investigator — Professor of Radiation Oncology
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place at Stanford University. The study started in July 2011 and it ended July 2014.
Pre-assignment Details: No pre-assignment details as the patients were recruited and placed directly in the study.
Groups:
- Intensity Modulated Radiotherapy Treatment: Radiation dose to the tumor is > 60 Gy at 1.8-2.2 Gy/fx.
  intensity modulated radiotherapy treatment
Period: Overall Study
Arm/Group | Intensity Modulated Radiotherapy Treatment
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intensity Modulated RT Treatment: Radiation dose to the tumor is > 60 Gy at 1.8-2.2 Gy/fx.
  intensity modulated radiotherapy treatment
Arm/Group | Intensity Modulated RT Treatment
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 61.5 [42 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 30
Primary Tumor location [Count of Participants; unit: Participants]
  Pharynx | 23
  Oral Cavity | 7
Tongue dose [Median (Full Range); unit: Gy] — Measurement of the lateral tongue mucosal dose was performed using optically stimulated luminescence (OSL) dosimeters, which were taped on the lingual side of the lower mouth-bite. The OSL was placed on the first day of RT in the 2 mucosal sites: lateral oral tongue on the left (L) and right (R) sides adjacent to dental fillings. The OSL was developed and measured on the same day. The measured dose per fraction was converted to the total dose for the entire treatment.
  Gy | 30.5 [11.2 to 70]

OUTCOME MEASURES:

1. Primary Outcome: Time Until the Maximum Oral Mucositis Measured From the Start of Radiation Treatment.
Description: The time to onset of oral mucositis was measured from the start of radiation treatment until oral mucositis was visual observed by a clinician during the weekly checkup for the first time. Analysis done by Kaplan-Meier.
  Adverse events were graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version (V) 4.0. Medical doctor performed evaluation and grading of clinical and functional mucositis for the measured site weekly during the radiation treatment course and biweekly after completion of radiation until oral mucositis was < grade 2. A pain medication assessment was done for each mucositis time point. Patients completed the Oral Mucositis Weekly Questionnaire-Head and Neck cancer (OMWQ-HN) during and after treatment until oral mucositis is < grade 2.
Time Frame: 3 years
Population: The entire cohort was analyzed
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Intensity Modulated Radiotherapy Treatment
Number analyzed (Participants) | 30
Days
  Dose <30 Gy | 34 [28 to 36]
  Dose >= 30 Gy | 29 [21 to 35]
Statistical Analysis 1: Comparison: Intensity Modulated Radiotherapy Treatment; Test type: Superiority or Other; p = 0.9906, Regression, Cox; This was a Cox proportional hazards model with dose as the single predictor; Cox Proportional Hazard = 1.000, 95% CI 2-sided [0.979 to 1.022]

2. Primary Outcome: Duration of Grade 2 or Higher Oral Mucositis After First Oral Mucositis Was Observed.
Description: The duration of grade 2 or higher oral mucositis was measured as the time from the first time oral mucositis was observed by a clinician at the weekly checkup until the oral mucositis was resolved.
  The data was analyzed in a mixed effects model to account for the within subject correlation, since each patient contributed two measurements to the data set. The model was limited to those subjects who had experienced mucositis and then the outcome was the duration of grade 2 or higher mucositis. This allowed us to model the data in a mixed effects model with the continuous outcome of duration of grade 2 or higher mucositis.
Time Frame: 3 years
Population: For each subject, both left and right sides were included as two measurements from the same individual.
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Intensity Modulated Radiotherapy Treatment
Number analyzed (Participants) | 25
Days
  dose < 30 Gy | 25.722 [14.692 to 36.752]
  dose >= 30 Gy | 27.917 [18.364 to 37.469]
Statistical Analysis 1: Comparison: Intensity Modulated Radiotherapy Treatment; Test type: Superiority or Other; p = 0.1209, Regression, Linear; Linear regression model with dose as the single predictor in the model; Slope = 0.2795, 95% CI 2-sided [-0.077 to 0.634]

3. Secondary Outcome: Relationship Between the Measured Lateral Tongue Mucosal Dose and the Amount of Narcotic Use
Description: The narcotics use was a patient reported measurement that was documented in the medical note in the patient chart. Patient self reported measurements are generally known to be unreliable.
Time Frame: 3 years
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Intensity Modulated Radiotherapy Treatment
Number analyzed (Participants) | 30
mg
  dose < 30 Gy | 917.5 [232.2 to 1602.8]
  dose >= 30 Gy | 1214.3 [552.2 to 1876.3]
Statistical Analysis 1: Comparison: Intensity Modulated Radiotherapy Treatment; Test type: Superiority or Other; p = 0.9832, Regression, Linear; Linear regression model with dose as the single predictor in the model; Slope = -0.285, 95% CI 2-sided [-27.28 to 26.71]

4. Secondary Outcome: How Does Increase in Soreness Scores Affect Quality of Life Questionnaire While Adjusting for the Measured Lateral Tongue Mucosal Dose
Description: The quality of life questionnaire was the HNC adaptation of the Oral Mucositis Daily Questionnaire (OMWQ). It is designed to assess the severity and impact of the oral mucositis by evaluating mouth and throat soreness and the degree to which the mouth and throat soreness interferes with activities of daily life such as eating, swallowing, drinking, talking and sleeping.
  This outcome measures soreness in both the mouth and throat.
  This outcome is not a combination of several sub-scales. This outcome was the response to the single question: "On a scale from 0 to 10, how would you rate your OVERALL MOUTH AND THROAT SORENESS during the past 24 hours?"
  Mouth and throat soreness was measured as a single scale from 0 (no soreness) to 10 (worst soreness possible).
Time Frame: 3 years
Measure: Mean (95% Confidence Interval); unit: units on soreness scale
Arm/Group | Intensity Modulated Radiotherapy Treatment
Number analyzed (Participants) | 30
units on soreness scale
  dose < 30 Gy | 2.908 [2.011 to 3.805]
  dose >= 30 Gy | 3.689 [2.832 to 4.546]
Statistical Analysis 1: Comparison: Intensity Modulated Radiotherapy Treatment; Test type: Superiority or Other; p = 0.0263, Mixed Models Analysis; A repeated measures model with dose as the single predictor. QoL values were measured for each patient every week; Slope = 0.03795, 95% CI 2-sided [0.00483 to 0.071]

5. Secondary Outcome: How Does Increase in Pain Scores Affect Quality of Life Questionnaire While Adjusting for the Measured Lateral Tongue Mucosal Dose?
Description: The quality of life questionnaire was the HNC adaptation of the Oral Mucositis Daily Questionnaire (OMDQ). It is designed to assess the severity and impact of the oral mucositis by evaluating mouth and throat soreness and the degree to which the mouth and throat soreness interferes with activities of daily life such as eating, swallowing, drinking, talking and sleeping.
  This outcome measures pain in the mouth only.
  This outcome is not a combination of several sub-scales. This outcome was the response to a single question: "On a scale from 0 to 10, what number best describes the MOUTH PAIN that you experienced in the past 24 hours?"
  Mouth pain scale was measured as a single scale from 0 (no pain) to 10 (worst pain imaginable).
Time Frame: 3 years
Population: Only 29 out of the 30 subjects filled out the pain surveys
Measure: Mean (95% Confidence Interval); unit: units on pain scale
Arm/Group | Intensity Modulated Radiotherapy Treatment
Number analyzed (Participants) | 29
units on pain scale
  dose < 30 Gy | 2.28 [1.278 to 3.283]
  dose >= 30 Gy | 3.292 [2.332 to 4.253]
Statistical Analysis 1: Comparison: Intensity Modulated Radiotherapy Treatment; Test type: Superiority or Other; p = 0.0039, Mixed Models Analysis; A repeated measures model with dose as the single predictor and QoL values measured each week for each patient; Slope = 0.0567, 95% CI 2-sided [0.0199 to 0.0935]

ADVERSE EVENTS:
Time Frame: The adverse events data was collected during the entire study period from July 2011 until July 2014 for a total of 3 years.
Arm/Group | Intensity Modulated Radiotherapy Treatment
Serious Adverse Events (participants affected / at risk) | 11/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensity Modulated Radiotherapy Treatment (N=30)
Mucositis Oral (Gastrointestinal disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No